CLINICAL TRIAL: NCT06329895
Title: A Phase 1, Open Label, Fixed Sequence, Crossover Study to Investigate the Effect of BAY 2927088 on the Pharmacokinetics of Dabigatran Etexilate or Rosuvastatin in Healthy Participants
Brief Title: A Study to Learn About How BAY2927088 Affects the Level of Dabigatran or Rosuvastatin in the Blood When These Drugs Are Taken Together in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 22252
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Advanced Non-small Cell Lung Cancer; EGFR Mutation; HER2 Mutation; Healthy Volunteers
Keywords: HER2; EGFR; NSCLC
MeSH Terms: interventions — Dabigatran; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): The healthy volunteers will be confined to the clinic throughout the Intervention Period of the study.
  The study includes visits during Screening, Intervention, and Follow-up.
  Interventions: Drug: BAY2927088; Drug: Dabigatran etexilate; Drug: Rosuvastatin

INTERVENTIONS:
Drug: BAY2927088 — Oral administration.
Drug: Dabigatran etexilate — Oral administration.
Drug: Rosuvastatin — Oral administration.

SUMMARY:
Researchers are looking for a better way to treat people who have advanced non-small cell lung cancer (NSCLC) with specific genetic changes called epidermal growth factor receptor (EGFR) and human epidermal growth factor receptor 2 (HER2) mutations.

Advanced NSCLC refers to a type of lung cancer that has spread from the lungs to nearby tissues or other body parts. People with advanced NSCLC may have changes in certain proteins, like EGFR and HER2, that cause uncontrolled cell growth and increased spread of cancer.

In this study, participants will be healthy and will not benefit from taking the study treatment, BAY2927088. However, the study will provide information about how to test BAY2927088 in future studies with people who have advanced NSCLC with EGFR or HER2 mutations.

BAY2927088 is under development for the treatment of advanced NSCLC with EGFR or HER2 mutations. It is expected to work against these changed proteins, which might slow down the spread of cancer.

Researchers think that BAY2927088 inhibits drug transporters such as P-gp (P-glycoprotein) and breast cancer resistance protein (BCRP). Drug transporters are proteins that help in the movement of certain drugs into, through, and out of the body's cells. Dabigatran is a drug used in the treatment of blood clots in a vein and rosuvastatin is a drug used in the treatment of high cholesterol in the blood.

The main purpose of this study is to find out how BAY2927088, taken as multiple doses, affects the levels of dabigatran and rosuvastatin in the blood of healthy participants. For this, researchers will measure the following for dabigatran and rosuvastatin, when given with and without BAY2927088:

* Area under the curve (AUC): a measure of the total amount of the drug in participants' blood over time
* Maximum observed concentration (Cmax): the highest amount of the drug in participants' blood

In this study, participants will take the following treatments:

* Dabigatran in the morning of Day 1 and 9.
* Rosuvastatin in the morning of Day 3 and 12.
* BAY2927088 two times a day in the morning and evening of Days 6 to 15.

Participants will be in this study for about 8 weeks with 3 visits to the study clinic.

Participants will visit the study clinic:

* at least once, 2 to 28 days before the treatment starts, to confirm they can take part in this study
* once on the day before the treatment starts and will stay in the clinic until Day 16 of the treatment
* once, 7 to 10 days after last dose of BAY2927088, for a health check-up

During the study, the doctors and their study team will:

* do physical examinations
* collect blood samples from the participants to measure the levels of dabigatran, rosuvastatin and of BAY2927088
* check participants' health by performing tests such as blood and urine tests, and checking heart health using an electrocardiogram (ECG)
* ask the participants questions about how they are feeling and what adverse events they are having

An adverse event is any medical problem that a participant has during a study. The study doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent as described in protocol which includes compliance with the requirements and restrictions listed in the informed consent form (ICF), and in this protocol.
* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by the investigator or medically qualified designee based on medical evaluation including medical history, laboratory tests, physical, and cardiac examination.
* Participant is a nonsmoker who has not used tobacco- or nicotine- containing products (e.g., nicotine patch) for at least 6 months before administration of the first study intervention.
* Body mass index (BMI) within the range 18.0 to 30 kg/m^2 (inclusive) at screening, with bodyweight above/equal to 50 kg.
* Female, of non-childbearing potential only

  * Females must not be pregnant or breastfeeding and must be documented as a woman of nonchildbearing potential. A negative pregnancy test is required.
  * Male study participants of reproductive potential must agree to use adequate contraception when sexually active.
* From signing of the ICF until at least 3 months after the last dose of study intervention, and refrain from sperm donation during study intervention and for 6 months after the last dose of study intervention.
* Participant must be willing to comply with dietary and fluid requirements during the study period (including abstaining from alcohol use).

Exclusion Criteria:

* Existing relevant diseases of vital organs (e.g., liver diseases, heart diseases, gastrointestinal diseases, interstitial lung disease, renal diseases), central nervous system (for example seizures) or other organs (e.g., diabetes mellitus).
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study intervention will not be normal.
* Febrile illness within 4 weeks prior to admission to the clinic.
* Any relevant diseases within 4 weeks prior to the first study intervention administration as judged by the investigator.
* A medical history of risk factors for Torsades de pointes (e.g., family history of long QT syndrome) or other clinically significant arrhythmias as judged by the investigator.
* Known severe allergies, allergies requiring therapy with corticosteroids, significant non-allergic drug reactions, or (multiple) drug allergies (excluding seasonal allergies such as non-severe hay fever that are asymptomatic and untreated during the time of study conduct).
* Known history of hypersensitivity (or known allergic reaction) to BAY 2927088-related compounds, or any components of the formulation, dabigatran etexilate or rosuvastatin.
* History of known or suspected malignant tumors.
* Participants who in the investigator's judgment are perceived as having an increased risk of bleeding.
* Known or suspected coagulopathies.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Cmax of unconjugated dabigatran when given with and without BAY2927088 | Pre-dose on Day 1 and 9, multiple post-dose time points on Day 1-2 and Day 9-11 and one time point on Day 3 and Day 12
  Cmax: Maximum observed drug concentration
AUC of unconjugated dabigatran when given with and without BAY2927088 | Pre-dose on Day 1 and 9, multiple post-dose time points on Day 1-2 and Day 9-11 and one time point on Day 3 and Day 12
  AUC: Area under the concentration vs time curve
Cmax of rosuvastatin when given with and without BAY2927088 | Pre-dose on Day 3, Day 12, multiple timepoints on Day 3-5, Day 12-15, one timepoint on Day 6 and Day 16
AUC of rosuvastatin when given with and without BAY2927088 | Pre-dose on Day 3, Day 12, multiple timepoints on Day 3-5, Day 12-15, one timepoint on Day 6 and Day 16

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 7 days after the last administration of study intervention
Severity of TEAEs | Up to 7 days after the last administration of study intervention

CONTACTS AND LOCATIONS:
Locations (1):
- PAREXEL International Early Phase Clinical Unit (London), Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/22252